CLINICAL TRIAL: NCT02544334
Title: Oral Metagenomic Biomarkers in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Medical Center-Gainesville (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB201500286; 11712325 (Other Grant/Funding Number: Department of Defense); 12.420 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2015-08-31; First posted 2015-09-09 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Metagenome; microbiome
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Dental Plaque Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Supragingival dental plaque will be pooled from different tooth surfaces using sterile periodontal curettes. DNA samples will be subjected to deep sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RA - naïve to biologics: This group will consist of 25 Rheumatoid Arthritis (RA) adult subjects who have not been treated with biologics (naïve to biologics). During the exam the following will take place: the multidimensional health assessment questionnaire (MDHAQ), dental exam, saliva collection, and dental plaque will be removed from different tooth surfaces for supragingival.
  Interventions: Procedure: Dental Plaque; Other: Multi-dimensional health assessment questionnaire (MDHAQ); Other: Saliva Collection
- Healthy Controls: This group will consist of 25 adult subjects which will be healthy controls from members of the same household as the 25 naive to biologics, and be of the same age. During the exam the following will take place: dental exam, saliva collection, and dental plaque will be removed from different tooth surfaces for supragingival.
  Interventions: Procedure: Dental Plaque; Other: Saliva Collection
- RA responsive to anti-TNF: This group will consist of 25 adult subjects with Rheumatoid Arthritis (RA) who have been responsive to first line anti-TNF-alpha therapy. During the exam the following will take place: the multidimensional health assessment questionnaire (MDHAQ), dental exam, saliva collection, and dental plaque will be removed from different tooth surfaces for supragingival.
  Interventions: Procedure: Dental Plaque; Other: Multi-dimensional health assessment questionnaire (MDHAQ); Other: Saliva Collection
- RA non responsive to anti-TNF: This group will consist of 25 adult subjects with Rheumatoid Arthritis (RA) who are resistant to two or more anti-TNF-alpha therapies, and be of the same age as the RA responsive to anti-TNF group. During the exam the following will take place: the multidimensional health assessment questionnaire (MDHAQ), dental exam, saliva collection, and dental plaque will be removed from different tooth surfaces for supragingival.
  Interventions: Procedure: Dental Plaque; Other: Multi-dimensional health assessment questionnaire (MDHAQ); Other: Saliva Collection

INTERVENTIONS:
Procedure: Dental Plaque — All participants will have dental plaque removed from different tooth surfaces for supragingival.
Other: Multi-dimensional health assessment questionnaire (MDHAQ) — The RA groups will receive the multi-dimensional health assessment questionnaire (MDHAQ) for physical function, pain, and global status.
  Other Names: MDHAQ
  Groups: RA - naïve to biologics; RA non responsive to anti-TNF; RA responsive to anti-TNF
Other: Saliva Collection — All participants will have a saliva collection.

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic and potentially severe autoimmune disease affecting 2 million in the United States. The role of environmental factors in modulating autoimmunity pathogenesis has been clearly described and yet the specific mechanisms of action remain poorly understood. A growing body of evidence implicates microbiota of mucosal surfaces in the development of autoimmune disorders. Various studies have clearly linked RA to periodontal disease. The latter is linked to the red-complex that includes the oral bacterium Porphyromonas gingivalis. And yet there has not been a systematic analysis of the oral microbiota in RA to determine whether there are specific markers for P. gingivalis (and other oral bacteria) that are linked to RA.

In this study, the investigators will characterize oral microbial composition (microbiome) and gene content (metagenome) of DNA isolated from oral samples obtained from patients with (i) early stage RA prior to biologics treatments and (ii) subsets of RA patients who are responsive or unresponsive to anti-TNF-alpha therapy. The innovative aspect of this study is going beyond the identification of oral bacterial species, to the level of strains and genes that are associated with these groups. The overall hypothesis is that oral microbial variation exists between individuals that influences development of autoimmunity and autoimmune disease.

DETAILED DESCRIPTION:
This is a multi-disciplinary research study with five investigators from different, yet complementary, disciplines to establish this new collaboration. There is a high translational potential for information gained from this project based on the collaboration of a rheumatologist, a dentist, oral biologists, and infectious disease experts with expertise in immunology, microbiology, and genomics. In brief, RA participants will be recruited by the rheumatologist. A total of 100 participants will be recruited for two groups to be studied; one group of subjects with RA and the other group will be healthy controls. These two groups will be divided into the following groups for participation in the study: Group 1: will consist of 25 RA adult subjects who have not been treated with biologics which will be compared to 25 healthy controls from age-matched members of the same household. Group 2 will consist of 25 RA adult subjects responsive to first line anti-TNF therapy which will be compared to 25 subjects of the same age and sex with RA who are resistant to two or more TNF antagonists. The participants will be scheduled for a research study visit at the University of Florida Dental Clinic Research Unit. During the exam the following will take place: the multidimensional health assessment questionnaire (MDHAQ), dental exam, saliva collection, and dental plaque will be removed from different tooth surfaces for supragingival.

The supragingival will be subjected to deep sequencing in the genomics lab. To test two specific aims: 1) testing the hypothesis that oral microbiome profiles based on 16S RNA data are associated with the development of RA or with the response to a specific therapy, and 2) testing the hypothesis that the specific genes, variants, and functional capabilities (metagenome) are associated with RA or with therapeutic response. Upon completion of this pilot study, the investigators will have systematically identified bacterial biomarkers (e.g. species, subspecies, genes) that correlate with RA and may serve as potential targets for disease treatment. These markers may be developed into new drug targets for RA therapy in future studies.

ELIGIBILITY:
Inclusion Criteria:

* with at least 10 natural uncrowned teeth (excluding third molars) must be present.

Exclusion Criteria:

* have less than 10 teeth;
* have been treated with antibiotics within the past 3 months, including patients that require antibiotic prophylaxis prior to dental treatment;
* are immune compromised individuals (HIV, AIDS, immuno-suppressive drug therapy);
* participate in another clinical study involving the use of dental products one week prior to the start of the washout period or during the study period; and
* are unwilling or unable to provide informed consent and follow the collection instructions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis (RA) adult patients who have not been treated with biologics (naïve to biologics), RA patients responsive to first line anti-TNF therapy, RA patients who are resistant to two or more TNF antagonists, and healthy controls from age-matched members of the same household.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-05; Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Oral microbiome will be catalogued in each group for their association with RA. | Day 1
  A Wilcoxon rank-sum test will be computed on each profile to identify differential metagenomic gene content between each pair of groups (RA patients and controls). The potential microbial functional roles of the KEGG orthologues and eggnog orthologue groups markers in the oral microbiota of RA patients will also be assessed. All results will be corrected for multiple testing using a false discovery rate approach.
Metagenomic analyses will be performed to find oral bacteria markers between the groups. | 18 months
  A Wilcoxon rank-sum test will be computed on each profile to identify differential metagenomic gene content between each groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Bubb, MD, Principal Investigator — University of Florida; Edward K Chan, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida College of Dentistry-Periodontics, Gainesville, Florida
  - Randall Malcom VA Medical Center, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided